CLINICAL TRIAL: NCT02233114
Title: Subjective and Objective Effects After Yogic Exercises
Brief Title: Is Patients With Pulmonary Disease Benefit a Program With Yogic Exercises?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Wandell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DNR2011/248-31/1
Record Dates: First submitted 2014-08-25; First posted 2014-09-08 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-09

CONDITIONS: COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yogic exercises (Experimental): Yogic exercises for lung disorders
  Interventions: Other: Yogic exercises
- physiotherapy (Active Comparator): Physiotherapy during the yogic exercises
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Yogic exercises — Yogic exercises (YE) - 2 hours per week, 1h in each session
  Arms: Yogic exercises
Other: Physiotherapy — Physiotherapy (low intensity cardiovascular training and strength training) - 2 hours per week, 1 h in each session
  Arms: physiotherapy

SUMMARY:
Is Yogic Exercises (12 weeks) increasing respiratory function, functional capacity and quality of life in patients with obstructive lung diseases. With follow up after 6 months.

DETAILED DESCRIPTION:
Is Yogic Exercises increasing respiratory function in patients with obstructive lung diseases. Will YE improve respiratory muscle strength, functional capacity, inspiratory and expiratory pressure, lung function, perceived dyspnea, dyspnea-related distress (DD), less frequency of dyspnea and heart rate variability in patients with pulmonary disease. Qualitative content analysis will be performed on approximately 15 interviews with patients participated in the yoga group about their experiences and their benefits perceived/experienced of the yogic exercises

We want to try YE as an alternative treatment in patients with mild to severe pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to severe pulmonary obstructions according to GOLD 1-3 (Global Initiative for Chronic Obstructive Lung Disease),
* FEV (forced expiratory volume) in one second (FEV1) % of predicted respiratory function (30% ≤ FEV1 ≤ 90%)
* FEV1/FVC < 0.70 (<65 over 65 yrs). *FVC=forced vital capacity

Exclusion Criteria:

* Severe neurological, orthopedic or rheumatologic injuries
* Severely decreased thorax mobility and lung function.
* Severe lung diseases
* Other chronic diseases that will interfere with performance.
* Under 200 meters on the 6MWT
* Acute dyspnea
* Surgery within 6 months
* Medication affecting attention, sudden change of medication.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Dyspnea related distress (DD) | Patients will be followed 10-12 weeks, with follow-up after 6 months
Functional capacity | Patients will be followed 10-12 weeks, with follow-up after 6 months
  6 minutes Walking test

SECONDARY OUTCOMES:
Spirometry, Vital capacity | Patients will be followed 10-12 weeks, with follow-up after 6 months
Oxygen saturation (periphery) | Patients will be followed 10-12 weeks, with follow-up after 6 months
Respiration rate | Patients will be followed 10-12 weeks, with follow-up after 6 months
  Measured manually
CRQ, Chronic respiratory disease questionnaire | Patients will be followed 10-12 weeks, with follow-up after 6 months
VAS- scale - perceived health | Patients will be followed 10-12 weeks, with follow-up after 6 months
  Scoring between 0 (worst possible) and 10 (best possible)
Maximal inspiratory and maximal expiratory pressure | Patients will be followed 10-12 weeks, with follow-up after 6 months
Perceived stress | Patients will be followed 10-12 weeks, with follow-up after 6 months
  Will be measured using PSS-14 scale
Sleep quality | Patients will be followed 10-12 weeks, with follow-up after 6 months
  Measured with Pittsburgh sleep questionnaire index scale
Anxiety and depression | Patients will be followed 10-12 weeks, with follow-up after 6 months
  Measured with HADS-scale
Self rated health | Patients will be followed 10-12 weeks, with follow-up after 6 months
Subjective complaints (perceived symptoms) | Patients will be followed 10-12 weeks, with follow-up after 6 months
Blood pressure | Patients will be followed 10-12 weeks, with follow-up after 6 months
Weight and height | Patients will be followed 10-12 weeks, with follow-up after 6 months
Health behaviour | Patients will be followed 10-12 weeks, with follow-up after 6 months
  Measured with public health questionnaire (Folkhälsoenkäten in Swedish)
Exercise diary | Patients will be followed 10-12 weeks, with follow-up after 6 months
Spirometry, forced vital capacity (FVC) | Patients will be followed for 10-12 weeks, with follow-up after 6 months
Spirometry, Forced expiratory volume | Patients will be followed for 10-12 weeks, with follow-up after 6 months
Spirometry, Forced expiratory volume in one second (FEV1) | Patients will be followed for 10-12 weeks, with follow-up after 6 months
Spirometry, Ratio between forced expiratory volume in 1 second and forced vital capacity | Patients will be followed for 10-12 weeks, with follow-up after 6 months
Spirometry, peak expiratory flow (PEF) | Patients will be followed for 10-12 weeks, with follow-up after 6 months
Insomnia | Patients will be followed for 10-12 weeks, with follow-up after 6 months
  Measured with insomnia index scale
Heart rate variability | Patients will be followed for 10-12 weeks, with follow-up after 6 months
  Measured with Polar heart rate monitor
Qualitative content analysis | After Yoga intervention - one interview, with follow-up after 6 months
  Inteviews with participants in yoga Group, and at follow-up also physiotherapy group

CONTACTS AND LOCATIONS:
Overall Officials: Per Wändell, MD, PhD, Principal Investigator — Karolinska Institutet, Stockholm
Locations (1):
- Karolinska University hospital, Stockholm, Huddinge, Sweden

REFERENCES:
- [Derived] Papp ME, Henriques M, Biguet G, Wandell PE, Nygren-Bonnier M. Experiences of hatha yogic exercises among patients with obstructive pulmonary diseases: A qualitative study. J Bodyw Mov Ther. 2018 Oct;22(4):896-903. doi: 10.1016/j.jbmt.2017.11.001. Epub 2017 Nov 8. PMID 30368332